CLINICAL TRIAL: NCT00326261
Title: Randomized Controlled Trial of Ultrasound Guided Needle Placement Versus Nerve Stimulation for Coracoid Infraclavicular Brachial Plexus Block
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Canadian Anesthesiologists' Society (Other)
Other Study IDs: 03-0126-AE
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2006-04

CONDITIONS: Patients Undergoing Hand Surgery
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Ultrasound compared to dual-endpoint nerve stimulator guided approach.
Procedure: Ultrasound

SUMMARY:
Nerve blocks for arm and hand surgery provide many advantages for patients including excellent pain control and reduction in general anesthesia-related adverse effects. Infraclavicular block is possibly the best method for performing regional anesthesia of the arm because of the consistent anesthesia of the whole arm and low incidence of serious adverse effects. Normally the anesthetist uses nerve stimulation to identify nerves supplying the forearm and hand. Recent research has indicated that to improve success from 60% to 79% two types of muscle stimulation must be sought before injection of local anesthetic. This can be time consuming, requires a significant learning process, increases complications and leaves 21% of patients with inadequate anesthesia requiring supplementation or general anesthesia. More recently practitioners have been using ultrasound imaging to direct the needle and watch local anesthetic spread around the nerves. Preliminary reports have documented that this technique is associated with much greater success than the nerve stimulation method. However a good quality study comparing the dual-endpoint infraclavicular technique with an ultrasound-guided technique has not been performed. This randomized study aims to rectify this deficiency by determining if ultrasound-guided infraclavicular block has a significantly greater success than the current standard, dual end-endpoint nerve stimulation technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective upper limb surgery at or below the elbow.
* Patients aged > 18 and < 80 years.
* ASA I-III.
* BMI < 35.

Exclusion Criteria:

* Inability to read, write or speak English. (This is necessary because subjects will have to follow detailed instructions to allow testing of motor and sensory function. it is not feasible to have an interpreter present in the block room during performance of these procedures).
* Contraindication to brachial plexus block.
* Existing neurological deficit in the area to be blocked.
* Known loco-regional malignancy or infection.
* Coagulopathy.
* Allergy to local anesthetic agents.
* Chest or shoulder deformities.
* Severe respiratory disease.
* Healed but dislocated clavicle fracture.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Colin JL McCartney, MBChB FRCA FCARCSI FRCPC, Principal Investigator — University Health Network, Toronto Western Hospital
Locations (1):
- University Health Network, Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Brull R, Lupu M, Perlas A, Chan VW, McCartney CJ. Compared with dual nerve stimulation, ultrasound guidance shortens the time for infraclavicular block performance. Can J Anaesth. 2009 Nov;56(11):812-8. doi: 10.1007/s12630-009-9170-2. PMID 19728002